CLINICAL TRIAL: NCT03590210
Title: NiTraSarc Combined Treatment With Nivolumab and Trabectedin in Patients With Metastatic or Inoperable Soft Tissue Sarcomas - The NiTraSarc Phase II Trial
Brief Title: Combined Treatment With Nivolumab and Trabectedin in Patients With Metastatic or Inoperable Soft Tissue Sarcomas
Acronym: NiTraSarc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); PharmaMar (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GISG-15; 2017-001083-38 (EudraCT Number)
Record Dates: First submitted 2018-06-21; First posted 2018-07-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Nivolumab

STUDY DESIGN:
Intervention Model Description: Two group, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - L-sarcoma (Experimental): Patients with unresectable or metastatic liposarcoma or leiomyosarcoma who received a prior anthracycline-containing regimen will receive drug treatment with trabectedin (1 cycle mono-therapy) followed by trabectedin/nivolumab combination (up to 15 additional cycles); 16 cycles in total
  Interventions: Drug: Trabectedin; Drug: Nivolumab
- Group B - non-L-sarcoma (Experimental): Patients with unresectable or metastatic soft tissue sarcoma other than liposarcoma or leiomyosarcoma who received a prior anthracycline-containing regimen (GIST excluded) will receive drug treatment with trabectedin (1 cycle mono-therapy) followed by trabectedin/nivolumab combination (up to 15 additional cycles); 16 cycles in total
  Interventions: Drug: Trabectedin; Drug: Nivolumab

INTERVENTIONS:
Drug: Trabectedin — Cycle 1 to 16 1.5mg/m² IV over 24 hours, q3w
  Other Names: Yondelis
Drug: Nivolumab — Cycle 2 to 16 240 mg IV over 30 minutes, q3w
  Other Names: Opdivo

SUMMARY:
The "NiTraSarc" trial evaluates the efficacy and feasibility (as determined by the safety and tolerability) of combined treatment with trabectedin and nivolumab in patients with metastatic or inoperable soft tissue sarcomas

DETAILED DESCRIPTION:
Undoubtedly, there is a strong medical need for new efficacious therapies for patients with advanced soft tissue sarcomas. While immune oncology treatment approaches like inhibition of immune checkpoints by administration of anti PD-1 / PD-L1 antibodies displayed very promising clinical activity in several types of tumors, current data points out to only limited activity of mono-agent immunotherapy in soft tissue sarcomas (especially in leiomyosarcomas) - although this type of tumor demonstrably displays a certain grade of immunogenicity. That means, STS patients are currently not able to benefit from the advancements in cancer immunotherapy which led to remarkable improvements in outcome in some other tumor entities in the last few years.

Interestingly, most recent data indicates that trabectedin could enhance the activity of immune-modulating agents via its influence on the tumor micro-environment and the reduction of tumor associated macrophages. Furthermore, first clinical data obtained from a feasibility study on combined nivolumab/trabectedin therapy in STS patients did not report on significant toxicities when combining the two agents, thereby justifying combination of nivolumab and trabectedin utilizing standard dosages.

Therefore, this phase II study will examine if combination of nivolumab with trabectedin is feasible (safe and well tolerated) and efficacious by utilizing potential synergistic effects of both agents. In the long run, the results of this phase II trial could build the basis for further evaluation of the efficacy of the trabectedin / nivolumab combination in a randomized clinical trial involving larger patient numbers. Finally, this could render patients with STS accessible to immunotherapeutics - a promising new class of drugs for anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

Group A:

1 Patients must have histologically confirmed liposarcoma or leiomyosarcoma

Group B:

1. Patients must have histologically confirmed soft tissue sarcoma (STS) other than liposarcoma or leiomyosarcoma (GIST excluded)

   Both Groups (A and B):
2. ≥ 1 prior systemic therapy for sarcoma, including adjuvant systemic therapy (anthracycline-containing regimen)
3. Signed Written Informed Consent
4. Men and women aged ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Measurable disease (according to RECIST criteria version 1.1)
7. Locally advanced/unresectable or metastatic disease
8. No prior therapy with ipilimumab or nivolumab, or any agent targeting programmed cell death 1 (PD-1), PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
9. No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation ≤ 28 days before study registration; no treatment with nitrosourea or mitomycin ≤ 42 days before study registration
10. Patients should have resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, version 4.0, grade 1 or less
11. Patients must have a formalin-fixed, paraffin-embedded (FFPE) tumor block OR 1 representative hematoxylin and eosin (H&E) and 20 unstained sarcoma tissue slides available for submission to central pathology review. If no archival tissue is available, a fresh biopsy has to be performed during screening.
12. Absolute neutrophil count (ANC) ≥ 1,500/mm3
13. Platelet count ≥ 100,000/mm3
14. Creatine phosphokinase (CPK) ≤2,5 x ULN
15. Creatinine ≤ 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance ≥ 60 mL/min (calculated by using the Cockcroft-Gault formula)
16. Total bilirubin ≤ upper limit of normal (ULN). If total bilirubin is greater than (>) ULN, measure indirect bilirubin to evaluate for Gilbert's syndrome (if direct bilirubin is within normal range, participant may be eligible).
17. AST/ALT ≤ 2.5 x upper limit of normal (ULN)
18. AP ≤ 2.5 x upper limit of normal (ULN)
19. Hemoglobin ≥ 9 g/dl. If hemoglobin <9 g/dl, blood transfusion is permitted. If hemoglobin cannot be enhanced to ≥ 9 g/dl, patient cannot be included into the study.
20. Thyroid stimulating hormone (TSH) within normal limits (WNL); supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH if free T4 is normal and patient is clinically euthyroid, patient is eligible
21. Not pregnant and not nursing; for women of childbearing potential who are sexually active, a negative pregnancy test (urinary or serum beta-HCG) at screening (performed ≤7 days prior to registration) is required.
22. Female participants must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (at the discretion of the investigator), or if sexually active, follow the contraceptive guidance in Appendix 4 throughout the duration of study treatment and for a minimum of 5 months after the last dose of study medication. Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm for a minimum of 7 months after the last dose of study medication.

Exclusion Criteria:

1. Prior exposure to trabectedin
2. Active known or suspected autoimmune disease (e.g. autoimmune colitis, autoimmune panhypopituitarism, autoimmune adrenal insufficiency)

   EXCEPT:

   i) Subjects with vitiligo, type 1 diabetes mellitus, resolved childhood asthma or atopy are permitted to enroll.

   ii) Subjects with suspected autoimmune thyroid disorders may be enrolled if they are currently euthyroid or with residual hypothyroidism requiring only hormone replacement.

   iii) Subjects with psoriasis requiring systemic therapy must be excluded from enrollment.
3. Patients with human immunodeficiency virus (HIV) infection are excluded unless cluster of differentiation (CD)4+ cells are > 350 and no viral load is detectable
4. Symptomatic, untreated, or uncontrolled brain metastases present
5. Known significant chronic liver disease, such as cirrhosis or active hepatitis B or C

   * Hepatitis B can be defined as (all of the following conditions must be met):

     * Hepatitis B surface antigen (HBsAg) > 6 months
     * Serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥2,000 IU/ml (104 copies/ml)
     * Persistent or intermittent elevation in alanine aminotransferase (ALT)/alanine aminotransferase (AST) levels
     * Liver biopsy showing chronic hepatitis with moderate or severe necroinflammation
   * Hepatitis C can be defined as:

     * Hepatitis C antibody (Ab) positive
     * Presence of hepatitis C virus (HCV) ribonucleic acid (RNA)
6. Known active pulmonary disease with hypoxia defined as:

   * Oxygen saturation < 85% on room air or
   * Oxygen saturation < 88% despite supplemental oxygen
7. Systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration
8. Myocardial infarct within 6 months before enrollment, New York Heart Association Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
9. Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension or diabetes, ongoing active infection, or psychiatric illness/social situation that may potentially impair the participant's compliance with study procedures
10. Unwilling or unable to have a central venous catheter
11. Known allergies, hypersensitivity, or intolerance to trabectedin, dexamethasone, or their excipients, or monoclonal antibodies (biologics) therapy
12. Pregnant or breast-feeding
13. Any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements
14. On-treatment participation in another clinical study in the period 30 days prior to start of study treatment and during the study.
15. History of allogeneic solid organ or tissue transplant including allogeneic hematopoetic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
progression free survival rate at 6 months - PFSR6 | after 6 months of treatment
  The primary efficacy endpoint of the trial is the progression-free survival rate after 6 months (PFSR6), assessed by applying RECIST 1.1.
safety, as measured by: - Incidence of adverse events (AEs), serious adverse events (SAEs), adverse events leading to discontinuation, and deaths - Incidence of clinical laboratory test abnormalities | through study completion, an average of 24 months
  The primary safety endpoint is to assess the feasibility of combined treatment with trabectedin and nivolumab in patients with metastatic or inoperable soft tissue sarcomas as determined by the safety and tolerability of the combination treatment.

SECONDARY OUTCOMES:
overall response rate (ORR) | through study completion, an average of 24 months
  Objective Response Rate (ORR) defined as the number and percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). Best overall response (BOR) is defined as the best response designation, recorded between the date of first dose and the date of the initial objectively documented tumor progression per RECIST v1.1 or the date of subsequent therapy or death date, whichever occurs first. For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination.
overall survival (OS) | through study completion, an average of 24 months
  OS is defined as the time from date of the first dosing date of any study medication to the date of death (due to any cause). Subjects who are alive will be censored at the last known alive dates.
progression-free survival (PFS) | through study completion, an average of 24 months
  PFS is defined as the time from the first dosing date of any study medication to the date of the first objectively documented tumor progression, as determined by investigators (per RECIST v1.1), or death due to any cause. Subjects who die without a reported prior progression will be considered to have progressed on the date of their death. Subjects who did not progress or die will be censored on the date of their last tumor assessment. Subjects who did not have any on study tumor assessments and did not die will be censored on the first dosing date of study medication. Subjects who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last tumor assessment prior to initiation of the subsequent anti-cancer therapy. In addition to PFS according to RECIST v1.1, PFS according to immune related RECIST 1.1 (irRECIST 1.1) will be determined.
duration of disease stabilization (DoDS) | through study completion, an average of 24 months
  Duration of disease stabilization is defined as the sum of duration of response (DoR) and duration of stable disease (DoS) in months. So DoDS is applicable to subjects with best overall response as either CR or PR or SD and it is defined as time from the first assessment of CR or PR or SD until the date of the first occurrence of PD, or until the date of death (if occurred within predefined time period). In case of censored event, the DoDS is censored on the date of last tumor assessment.
PDL-1 expression | through study completion, an average of 24 months
  PDL-1 expression will be quantified during central pathological examination

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pink, MD, Principal Investigator — Klinik und Poliklinik für Innere Medizin C, Hämatologie und Onkologie, Transplantationszentrum, Universitätsmedizin Greifswald
Locations (9):
- Germany (9):
  - Helios Klinikum Bad Saarow, Klinik für Hämatologie, Onkologie und Palliativmedizin, Sarkomzentrum Berlin-Brandenburg, Bad Saarow
  - Helios Klinikum Berlin Buch, Klinik für interdisziplinäre Onkologie, Sarkomzentrum Berlin-Brandenburg, Berlin
  - Charité Universitätsmedizin Berlin, Campus Virchow Klinikum Medizinische Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunologie (CC14), Berlin
  - Medizinische Fakultät "Carl Gustav Carus" der TU Dresden, Medizinische Klinik I, Dresden
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Innere Medizin C, Hämatologie und Onkologie, Greifswald
  - Universitätsklinikum Medizinische Fakultät Mannheim der Universität Heidelberg, Interdisziplinäres Tumorzentrum Mannheim (ITM), Mannheim
  - Universitätsklinikum Münster, Medizinische Klinik A Hämatologie / Onkologie / Pneumologie, Münster
  - Universitätsklinikum Tübingen, Innere Medizin II - Medizinische Onkologie und Pneumologie, Tübingen
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II Hämatologie / Onkologie, Würzburg

IPD SHARING:
Plan to Share IPD: No